CLINICAL TRIAL: NCT01685684
Title: A Phase 3, Multi-Center, Randomized, Double-blind, Placebo-Controlled, Safety, Tolerability, and Efficacy Study of Oxycodone DETERx™ Versus Placebo in Opioid-Experienced and Opioid-Naive Subjects With Moderate-to-Severe Chronic Low Back Pain
Brief Title: Oxycodone DETERx™ Versus Placebo in Chronic Low Back Pain (CLBP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Collegium Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-OXYDET-08
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-02

CONDITIONS: Chronic Low Back Pain
Keywords: Low back pain; Chronic back pain; Back pain; Opioid; Oxycodone; DETERx; Chronic pain; Chronic low back pain; CLBP; Xtampza
MeSH Terms: conditions — Low Back Pain; Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone DETERx (Experimental)
  Interventions: Drug: Oxycodone DETERx
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone DETERx — 40-160 mg total daily dose of oxycodone DETERx, divided into 2 doses, q12h
  Arms: Oxycodone DETERx
Drug: Placebo — Placebo, divided into 2 doses, q12h
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy of Oxycodone DETERx compared with placebo in opioid-experienced and opioid-naive subjects with moderate-to-severe chronic low back pain requiring around-the-clock opioid analgesia for an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female 18-75 years of age (inclusive) at the time of consent.
* Must have a clinical diagnosis of moderate-to-severe CLBP for a minimum of 6 months prior to screening.
* Must qualify for ATC opioid therapy for treatment of CLBP.
* Must be classified as non-malignant and non-neuropathic (Class 1 and 2), neuropathic (Class 3), or symptomatic for more than 6 months after low back pain surgery (Class 9) based on the Quebec Task Force Scale score.
* Female subjects of childbearing potential will use an acceptable method of birth control.
* Must be in general good health based on screening physical examination.
* Must be willing and able to comply with all study procedures and visit requirements.

Exclusion Criteria:

* Known to be refractory or intolerant to the analgesic effects of opioids or have failed previous opioid therapy.
* A medical condition that would compromise the subject's ability to swallow, absorb, metabolize, or excrete the study drug, including (but not limited to) intractable nausea and/or vomiting and/or severe gastrointestinal narrowing (pathologic or iatrogenic), bowel obstruction, ileostomy, colostomy, or is suspected of having paralytic ileus.
* A surgical procedure for back pain within 6 months prior to the Screening Visit.
* Any other chronic pain condition other than CLBP that would interfere with the assessment of CLBP (e.g., osteoarthritis, rheumatoid arthritis, post-herpetic neuralgia, pain associated with diabetic neuropathy, fibromyalgia, migraine headaches requiring opioid therapy).
* Known history of major depressive disorder that is not controlled with medication or has other conditions that produce significant cognitive or emotional disability.
* Any clinically significant unstable medical abnormality or acute or chronic disease of the cardiovascular, gastrointestinal, respiratory (e.g., chronic obstructive pulmonary disease), hepatic, or renal systems.
* Known history of alcohol and/or drug abuse.
* Positive urine drug screen for illegal or non-prescribed drugs
* Known history of seizure disorder, epilepsy, convulsions, or increased intracranial pressure anytime during the subject's life except pediatric febrile seizures.
* Known history of head injury within 6 months of Screening Visit.
* Current malignancy or a history within past 2 years of malignancy, with the exception of basal cell carcinoma or cervical carcinoma in situ that have been successfully treated.
* Positive for human immunodeficiency virus (HIV) or hepatitis B surface antigen, or hepatitis C antibody
* Subject is not able or is unwilling to meet the study attendance requirements.

Other protocol specific inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Malamut, MD, Study Director — Collegium Pharmaceutical, Inc.
Locations (44):
- United States (44):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Buena Park, California
  - Cerritos, California
  - Escondido, California
  - La Mesa, California
  - Napa, California
  - Pasadena, California
  - DeLand, Florida
  - Naples, Florida
  - Orlando, Florida
  - Plantation, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Valparaiso, Indiana
  - Overland Park, Kansas
  - Brockton, Massachusetts
  - Natick, Massachusetts
  - Watertown, Massachusetts
  - Pascagoula, Mississippi
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - New York, New York
  - Rochester, New York
  - Williamsville, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Rapid City, South Dakota
  - New Tazewell, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Roanoke, Virginia
  - Bellevue, Washington

REFERENCES:
- [Result] Katz N, Kopecky EA, O'Connor M, Brown RH, Fleming AB. A phase 3, multicenter, randomized, double-blind, placebo-controlled, safety, tolerability, and efficacy study of Xtampza ER in patients with moderate-to-severe chronic low back pain. Pain. 2015 Dec;156(12):2458-2467. doi: 10.1097/j.pain.0000000000000315. PMID 26262828
- [Derived] Kopecky EA, Vaughn B, Lagasse S, O'Connor M. Tolerability, Safety, and Effectiveness of Oxycodone DETERx in Elderly Patients >/=65 Years of Age with Chronic Low Back Pain: A Randomized Controlled Trial. Drugs Aging. 2017 Aug;34(8):603-613. doi: 10.1007/s40266-017-0473-7. PMID 28600725

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The titration (i.e., enrichment) phase of the study was designed to titrate patients to a dose of Oxycodone DETERx that balanced pain control and tolerability to ensure that only patients who experienced a substantial reduction from the screening pain assessment and who can tolerate side effects continue into the Double-blind Maintenance Phase.
Groups:
- Oxycodone DETERx (Titration Phase): Achieve a stable Oxycodone DETERx dose of 40-160 mg total daily dose.
- Oxycodone DETERx (Double-blind Maintenance Phase): Oxycodone DETERx: 40-160 mg total daily dose of oxycodone DETERx, divided into 2 doses, q12h
- Placebo (Double-blind Maintenance Phase): Placebo: Placebo, divided into 2 doses, q12h
Period: Titration Phase
Arm/Group | Oxycodone DETERx (Titration Phase) | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Started | 740 | 0 | 0
Completed | 389 | 0 | 0
Not Completed | 351 | 0 | 0
Period: Double-blind Maintenance Phase
Arm/Group | Oxycodone DETERx (Titration Phase) | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Started | 0 | 193 | 196
Completed | 0 | 122 | 100
Not Completed | 0 | 71 | 96

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase) | Total
Number analyzed (Participants) | 193 | 196 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.31) | 49.9 (12.56) | 49.5 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 103 | 206
  Male | 90 | 93 | 183
Pain Intensity-Numeric Rating Scale (PI-NRS) [Mean (Standard Deviation); unit: units on a scale] — The PI-NRS is an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain).
  units on a scale | 3.0 (1.04) | 2.9 (0.97) | 2.9 (1.00)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Pain Intensity Measured by the Change in Pain Intensity-Numeric Rating Scale (PI-NRS) Scores From Randomization Baseline to Week 12 of the Double-blind Maintenance Phase
Description: The PI-NRS is an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Randomized Baseline through Week 12
Population: One subject is missing all Average Weekly Pain Scores after Screening in the Oxycodone DETERx treatment group. This subject has been excluded from the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 192 | 196
units on a scale | 0.29 (0.146) | 1.85 (0.223)
Statistical Analysis 1: Comparison: Oxycodone DETERx (Double-blind Maintenance Phase) vs Placebo (Double-blind Maintenance Phase); Test type: Superiority or Other; p < 0.0001, z-test; Marginal Mean Difference (Net) = -1.56, Standard Error of Mean 0.267

2. Secondary Outcome: Time-to-exit From the Study for All Causes
Description: Survival analysis. Measure type indicated as 'Number' below represents 25% quartile, given that the median was not reached. These data are consistent with subject completion in the Participant Flow module.
Time Frame: Randomization Baseline through Week 12
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 193 | 196
Days | 58.0 [37.0 to 78.0] | 35.0 [29.0 to 38.0]

3. Secondary Outcome: Percent Reduction in Pain Intensity for Responders
Description: Includes the cumulative distribution of subjects with an improvement in pain intensity, as measured on an 11-point PI-NRS scale, and the proportion of responders with at least 30% and at least 50% reduction in pain intensity.
Time Frame: Screening Baseline through Week 12
Measure: Number; unit: participants
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 193 | 196
participants
  Subjects with 30% Improvement | 95 | 65
  Subjects with 50% Improvement | 74 | 48

4. Secondary Outcome: Weekly Changes in Pain Intensity
Description: Weekly pain intensity scores were calculated based on averaged daily pain intensity scores (PI-NRS). Increases to the weekly change in pain intensity, correspond to increases in the PI-NRS scores (i.e. more pain).
Time Frame: Randomization Baseline and weekly through Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 193 | 196
units on a scale
  Week 1 | 0.1 (0.85) | 0.3 (1.17)
  Week 2 | 0.0 (1.05) | 0.4 (1.46)
  Week 3 | 0.1 (1.14) | 0.5 (1.78)
  Week 4 | 0.1 (1.25) | 0.8 (1.86)
  Week 5 | 0.2 (1.41) | 0.7 (1.86)
  Week 6 | 0.2 (1.45) | 0.7 (1.95)
  Week 7 | 0.1 (1.35) | 0.7 (2.00)
  Week 8 | 0.0 (1.29) | 0.8 (2.06)
  Week 9 | 0.1 (1.59) | 0.7 (2.15)
  Week 10 | 0.2 (1.55) | 0.7 (2.20)
  Week 11 | 0.2 (1.62) | 0.8 (2.23)
  Week 12 | 0.3 (1.54) | 0.8 (2.29)

5. Secondary Outcome: Rescue Medication Usage by Dose
Description: Evaluation of the total amount of rescue medication used (number of doses per day, number of doses per week, and total number of doses while on-study)
Time Frame: Randomization Baseline through Week 12
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 193 | 196
doses
  Doses per Day | 0.15 (0.297) | 0.23 (0.458)
  Doses per Week | 1.04 (2.081) | 1.60 (3.206)
  Total Number of Doses | 8.0 (16.38) | 11.2 (31.55)

6. Secondary Outcome: Rescue Medication Use by Dosage
Description: Evaluation of the total amount of rescue medication used (by milligrams of dosage per day, dosage per week, and total dosage while on-study)
Time Frame: Randomization Baseline through Week 12
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 193 | 196
milligrams
  Dosage per Day | 144.63 (289.472) | 189.32 (317.605)
  Dosage per Week | 1012.39 (2026.298) | 1325.27 (2223.231)
  Total Dosage | 7873.1 (16665.70) | 9028.1 (20441.67)

7. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC scale is a self-reported assessment that assesses a subject's impression of his/her change in activity limitations, symptoms, emotions, and the overall quality of life as they relate to his/her painful condition. The 7-point PGIC assessment includes "very much improved", "improved", "a little improved", "no change", "a little worse", "worse", and "very much worse".
Time Frame: Screening Baseline through Week 12
Measure: Number; unit: participants
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 122 | 100
participants
  Very Much Improved | 36 | 17
  Improved | 52 | 39
  A Little Improved | 23 | 26
  No Change | 9 | 12
  A Little Worse | 0 | 4
  Worse | 2 | 1
  Very Much Worse | 0 | 1

8. Secondary Outcome: Changes in Quality of Life
Description: Short Form 12 Question Health Survey version 2 (SF-12v2) is a self-report survey designed to measure general quality of life from the subject's point of view. The survey includes eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Physical (PCS) and mental component scores (MCS) are also calculated. Positive values indicate improvement from randomization baseline to Week 12.
Time Frame: Randomization Baseline through Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 193 | 196
units on a scale
  Physical Component Score | 7.524 (10.1327) | 3.622 (9.4290)
  Mental Component Score | -2.554 (10.4145) | 0.674 (11.1676)
  Physical Functioning | 0.6 (1.35) | 0.5 (1.00)
  Role Physical | 1.2 (2.35) | 0.6 (2.16)
  Bodily Pain | 0.7 (1.16) | 0.4 (1.29)
  General Health | 0.28 (0.784) | 0.22 (0.789)

9. Secondary Outcome: Change in Level of Physical Disability Using the Roland Morris Disability Questionnaire (RMDQ)
Description: The Roland Morris Disability Questionnaire (RMDQ) is a self-administered questionnaire designed to assess physical disability caused by lower back pain. The RMDQ contains 24 sentences that subjects used to describe themselves when they have back pain. The RMDQ score is the total number of items checked which is from a minimum of 0 to a maximum of 24; the greater the score the grater the physical disability due to lower back pain.
Time Frame: Randomization Baseline and Week 12
Population: The RMDQ was analyzed and presented as a change from Randomization Baseline to Week 12. Subjects' scores from Early Discontinuation visits were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Number analyzed (Participants) | 109 | 90
units on a scale | 0.4 (4.83) | 0.7 (5.32)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of first dose with study drug to the End-of-Study Visit/Early Discontinuation Visit. All AEs that were ongoing at the subject's last study visit were to be followed until resolution or for 30 days after the subject's last study drug dose, whichever came first.
Description: Serious adverse events (SAEs) were collected from informed consent until 30 days post last dose. If the Investigator became aware of an SAE within 30 days after the subject's last study drug dose, or through the last study visit, the SAE was to be reported. All SAEs, including those ongoing at End-of-Study/Early Discontinuation, were followed until resolution or until the outcome became chronically stable, or if no additional information could be obtained after unsuccessful contact attempts.
Groups:
- Screening: Serious Adverse Event (SAE) collection started during screening.
Arm/Group | Screening | Oxycodone DETERx (Titration Phase) | Oxycodone DETERx (Double-blind Maintenance Phase) | Placebo (Double-blind Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 2/1297 | 8/740 | 2/193 | 2/196
Other Adverse Events (participants affected / at risk) | 0/0 | 531/740 | 60/193 | 39/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening (N=1297) | Oxycodone DETERx (Titration Phase) (N=740) | Oxycodone DETERx (Double-blind Maintenance Phase) (N=193) | Placebo (Double-blind Maintenance Phase) (N=196)
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0 — Not related to study drug as assessed by Principal Investigator and Medical Monitor
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Screening (N=0) | Oxycodone DETERx (Titration Phase) (N=740) | Oxycodone DETERx (Double-blind Maintenance Phase) (N=193) | Placebo (Double-blind Maintenance Phase) (N=196)
Nausea (Gastrointestinal disorders) | 0 | 123 | 21 | 9 — Non-serious Adverse Events were not collected during screening.
Headache (Nervous system disorders) | 0 | 103 | 12 | 23 — Non-serious Adverse Events were not collected during screening.
Constipation (Gastrointestinal disorders) | 0 | 96 | 10 | 1 — Non-serious Adverse Events were not collected during screening.
Somnolence (Nervous system disorders) | 0 | 65 | 1 | 0 — Non-serious Adverse Events were not collected during screening.
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 55 | 5 | 3 — Non-serious Adverse Events were not collected during screening.
Vomiting (Gastrointestinal disorders) | 0 | 47 | 8 | 3 — Non-serious Adverse Events were not collected during screening.
Dizziness (Nervous system disorders) | 0 | 42 | 3 | 0 — Non-serious Adverse Events were not collected during screening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a joint manuscript has not been submitted for publication within twelve (12) months of completion or termination of the study, the PI is free to publish separately, upon provision of any proposed publication or manuscript to the Sponsor at least sixty (60) days before it is submitted or otherwise disclosed.